CLINICAL TRIAL: NCT04210531
Title: Effects of Beetroot Juice Supplementation in Neuromuscular Performance and Match Activity in Young Basketball Players
Brief Title: Beetroot Juice Supplementation in Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Collaborators: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, Javier Courel Ibáñez, Principal Investigator, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2421/2019
Record Dates: First submitted 2019-12-19; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Dietary Supplement; Sport Performance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BJ supplementation (Experimental): Acute beetroot juice (BJ) supplementation
  Interventions: Dietary Supplement: Beetroot juice (BJ) acute supplementation
- PLA supplementation (Placebo Comparator): Acute placebo (PLA) supplementation
  Interventions: Dietary Supplement: Placebo acute supplementation

INTERVENTIONS:
Dietary Supplement: Beetroot juice (BJ) acute supplementation — One serving 140 mL of BJ (12.8 mmol of NO3-; Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) after an overnight fast and 3 h before initiating the testing session.
  Arms: BJ supplementation
Dietary Supplement: Placebo acute supplementation — One serving placebo drink (0.08 mmol of NO3-; Salud Viva, Nano Salud 32 S.L) after an overnight fast and 3 h before initiating the testing session.
  Arms: PLA supplementation

SUMMARY:
Whereas beetroot juice (BJ) supplementation is shown to increase physical performance in endurance activities, its benefits in team sports has been barely studied. In this randomized placebo-controlled study, we investigated the effects of BJ acute supplementation in improving neuromuscular performance and physical match activity in basketball.

DETAILED DESCRIPTION:
Whereas beetroot juice (BJ) supplementation is shown to increase physical performance in endurance activities, its benefits in team sports has been barely studied. In this randomized placebo-controlled study, we investigated the effects of BJ acute supplementation in improving neuromuscular performance and physical match activity in basketball.Testing sessions will comprised a neuromuscular test battery consisting of a countermovement jump (CMJ), isometric handgrip strength, 10-m/20-m sprint and agility T-test, followed by a 40-minute simulated basketball match. Physical match activity (distances, speeds, accelerations and decelerations) will be monitored in real time using an inertial tracking system

ELIGIBILITY:
Inclusion Criteria:

* active basketball player
* more than 5 years of basketball training experience

Exclusion Criteria:

* concurrently participating in other studies
* contraindications to BJ diet
* physical limitations, health problems, or musculoskeletal injuries

Ages: 15 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-06-09 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Changes in baskeball 5-on-5 game activity (m/min) | 1 week
  Using a wireless inertial movement unit system

SECONDARY OUTCOMES:
Changes in maximal isometric handgrip strength (kg) | 1 week
  Using a dynamometer
Changes in maximal jump height (cm) | 1 week
  Maximal jump height using a contact platform
Changes in sprint time (s) | 1 week
  Time to complete 10-m and 20-m sprints using photocell timing gates
Changes in agility test (s) | 1 week
  Time to complete the modified T-test using photocell timing gates

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport Sciences, Murcia, San Javier, Spain